CLINICAL TRIAL: NCT01454375
Title: Emergency Department Tobacco Cessation Counseling: Implementation and Evaluation of a Community-Based Program
Brief Title: Emergency Department Smoking Cessation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: H10-01625
Record Dates: First submitted 2011-10-15; First posted 2011-10-19 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Tobacco Use Cessation
Keywords: Smoking
MeSH Terms: conditions — Tobacco Use Cessation; Smoking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (No Intervention): No change in current practice
- Referral fo QuitNow Services (Experimental): Behavioural - referral to QuitNow Services, smoking cessation counseling telephone line supported by the Ministry of Healthy Living and Sport
  Interventions: Behavioral: Referral to QuitNow Services

INTERVENTIONS:
Behavioral: Referral to QuitNow Services — QuitNow Services is a telephone counseling program supported by the Ministry of Health Living and Sport that counsels individuals to stop smoking
  Arms: Referral fo QuitNow Services

SUMMARY:
Tobacco smoke claims approximately 6000 lives annually in BC. In this study, the investigators will determine whether referring smoking patients from the Vancouver General Hospital Emergency Department to the investigators provincial QuitNow smoking cessation service will lead to improved patient outcomes, including number of cigarettes smoked, any quit attempts, and actual smoking cessation.

Participants in the usual care arm will receive standard care. Participants in the intervention arm will be eligible for referral to QuitNow Services, where telephone counseling will be offered. Further follow-up on all enrolled patients will be conducted at 1, 3, 6, and 12 months to re-assess smoking status.

The investigators hypothesis is that the intervention arm will have a higher quit rate that the control arm.

DETAILED DESCRIPTION:
As the leading cause of preventable deaths in British Columbia (BC), tobacco smoke claims approximately 6000 lives annually in BC. Although 16% of British Columbians smoke, the prevalence of smoking may be as high as 48% in the Emergency Department (ED) patient population. In this study, the investigators will determine whether referring stable adult smoking patients from the Vancouver General Hospital ED directly to the investigators provincial QuitNow smoking cessation service will lead to improved patient outcomes, including number of cigarettes smoked, any quit attempts, and actual smoking cessation. This will be the first ever randomized controlled trial to determine whether smokers referred from the ED to a web and phone based community resource will receive benefit.

Currently, EDs in British Columbia, including VGH, are not routinely counseling patients to stop smoking. However, up to 44% of ED patients do not have a family practitioner and rely solely on EDs for their health care. Therefore, the ED serves as a critical venue where smoking cessation can be initiated or reinforced. The BC Ministry of Health has recently funded a program called QuitNow, which in collaboration with the BC Lung Association, offers smoking cessation advice through an internet resource and a 24-hour telephone quit line. This year, a meta-analysis of randomized controlled trials showed that web-based and computer-based smoking cessation programs led to a significant increase in patients who stopped smoking, with effects that were sustained at 12 months. However, these studies did not include ED patients.

In this trial, participants assigned to the usual care arm will receive standard care, with no additional study-related smoking cessation counseling. Participants assigned to the intervention arm will be eligible for referral to the QuitNow service. In the intervention arm, individuals will receive telephone follow-up from QuitNow at their earliest convenience. For all participants, data will be collected on demographic information, chief complaint, past medical history, smoking history, medications including nicotine replacement therapies, and final diagnosis. The smoking history will include the patient's number of daily cigarettes smoked, years of smoking, any previous quit attempts, and desire to quit. Further telephone follow-up on all enrolled patients will be conducted at 1, 3, 6, and 12 months to re-assess smoking status. We will also determine whether participants were enrolled in or completed the QuitNow Services program. For our initial pilot study, we made 5 calls to each participant at each follow-up period. For this full randomized controlled trial, participants will be called a maximum of 15 times at 12 months.

Data analysis will be performed using individual growth curve analyses with a multi-level regression model. P values of <0.05 will be considered statistically significant. An intention-to-treat analysis will be performed. If results are found to be significant, a Benjamini-Hochberg adjustment for multiple comparisons will be done. The expected time commitment for each patient will be 15 minutes in the ED and 20 minutes total for 4 follow-up telephone phone calls.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* stable (vital signs within normal limits not requiring immediate physician intervention)
* used a tobacco product in the last 30 days
* presenting to the Vancouver General Hospital Emergency Department
* can provide informed consent in English

Exclusion Criteria:

* cannot provide informed consent
* sexual assault patients
* not a resident of British Columbia
* unable to provide telephone number of email address for follow-up

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1301 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Smoking cessation rates between intervention and control arms | 12 months
  Smoking cessation rate between intervention and control arms at 12 months

SECONDARY OUTCOMES:
Smoking cessation rates between intervention and control arms | 1 month
Smoking cessation rates between intervention and control arms | 3 months
Smoking cessation rates between intervention and control arms | 6 months
No of cigarettes smoked daily between intervention and control arms | 1, 3, 6, and 12 months
Differences in readiness for change between the intervention and control arms | 1, 3, 6, and 12 months
Differences in knowledge and attitudes concerning smoking between the intervention and control arms | 1, 3, 6, and 12 months
Differences in use of nicotine replacement therapies between the intervention and control arms | 1, 3, 6, and 12 months
Differences in number of quit attempts between the intervention and control arms | 1,3,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wai Cheung, MD, MPH, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital Emergency Department, University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Tsai APY, Tsai JP, Stewart L, Brubacher J, Cheung KW. Prevalence of potential smoking-related conditions among tobacco users in the emergency department and their perception that their visit may be smoking-related. CJEM. 2017 May;19(3):207-212. doi: 10.1017/cem.2016.381. Epub 2016 Oct 17. PMID 27748218
- See also: QuitNow Services website — http://www.quitnow.ca/index.php